CLINICAL TRIAL: NCT03571581
Title: Exploring the Role of Mindfulness Training in the Promotion of Medication Adherence in Heart Failure Outpatients.
Brief Title: Mind Your Heart Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Elena Salmoirago-Blotcher, Research Scientist, The Miriam Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R21HL140492 (NIH); R21HL140492 (NIH)
Record Dates: First submitted 2018-06-05; First posted 2018-06-27 (Actual); Results first posted 2022-08-29 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2022-08

CONDITIONS: Medication Non-adherence
Keywords: Medication adherence; Heart failure; Mindfulness interventions
MeSH Terms: conditions — Medication Adherence; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness Training (MT) (Experimental): Eight, 30-minute phone delivered MT sessions once a week for 8 weeks
  Interventions: Behavioral: Mindfulness Training (MT)

INTERVENTIONS:
Behavioral: Mindfulness Training (MT) — Participants assigned to the MT condition will receive a phone-delivered 30-minute mindfulness training once a week for 8 weeks. In addition to the weekly training session, participants will be instructed to practice mindfulness techniques for 20 minutes daily using a standardized audio recording to guide the participant through the techniques learned with the instructor.

SUMMARY:
This study investigated the feasibility and acceptability of a phone-delivered mindfulness intervention to improve medication adherence among outpatients with heart failure.

DETAILED DESCRIPTION:
This project seeked to study the role of mindfulness training (MT) in the promotion of medication adherence among patients with chronic heart failure (HF). A prospective pre/post design study was conducted among 50 stable outpatients with HF and sub-optimal self-reported medication adherence. MT sessions (one 30-min session/week over 8 weeks) were phone-delivered by qualified mindfulness instructors. Assessments were conducted at baseline, 3 months (end of the intervention) and 6 months since baseline. The primary outcomes were feasibility and acceptability. We hypothesized we would meet recruitment goals (n=50) within the study timeline, with < 20% drop out rates by the end of the study and that > 80% of participants would report high (=grade 5) enjoyment ratings on a self-report intervention enjoyment scale (range:1 to 5). Secondary outcomes were self-reported and objectively assessed medication adherence and functional capacity (a clinical marker of medication adherence. We hypothesized we would observe significant pre-post intervention improvements in medication adherence and functional capacity. Additional outcomes included possible mediators of intervention effect, i.e., cognitive function, mood, sleep quality, and interoceptive awareness.

ELIGIBILITY:
Inclusion Criteria:

* Age > = 18
* Fluency in English language
* A confirmed diagnosis of heart failure
* Sub-optimal adherence to medications
* Access to a telephone
* Ability to understand and speak English

Exclusion Criteria:

* Unwillingness/inability to provide informed consent
* New York Heart Association (NYHA) class IV heart failure or clinically unstable
* Severe hearing impairment not allowing phone delivery
* Severe depressive symptoms
* Acute psychosis
* Severe cognitive impairment
* Recent hospitalization (< 6 weeks)
* Current (at least once a month) mind/body practice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elena Salmoirago-Blotcher, MD, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Data generated under the project will be shared as per the NIH Grant Policy and The Miriam Hospital IRB guidelines. De-identified research data will be made available in a timely manner once the main findings from the final research data set have been accepted for publication. Access to these data will be available for educational or research purposes. Data will be de-identified to avoid linkages to individual research participants and will not contain variables that could lead to the disclosure of the identity of individual subjects. All requestors will be asked to sign a data sharing agreement that includes conditions to 1) protect the identity of participants, 2) limit use of data for educational and research purposes, 3) prevent transfer of data to other users, and 4) acknowledge the data source. The de-identified data will be shared using Excel or SPSS file formats.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Once the main findings from the final research data set have been accepted for publication.
Access Criteria: Researchers interested in obtaining the de-identified data and associated documentation (e.g. codebook) can make a request to the principal investigator by email.

REFERENCES:
- [Background] Salmoirago-Blotcher E. A treatment in search of a disease? Challenges in mindfulness research and practice. Explore (NY). 2022 Sep-Oct;18(5):509-514. doi: 10.1016/j.explore.2021.05.005. Epub 2021 May 26. PMID 34099424
- [Result] Salmoirago-Blotcher E, Walaska K, Trivedi D, Dunsinger S, Levine D, Breault C, Wu JR, Bock B, Cohen R. Exploring effects of mindfulness training on medication adherence in patients with heart failure: THE MIND YOUR HEART STUDY. Annals of Behavioral Medicine. 2021; 55: S210-S210.
- [Result] Salmoirago-Blotcher E, Walaska K, Trivedi D, Dunsiger S, Levine D, Breault C, Wu JR, and Cohen R.Effects Of Mindfulness Training On Cognitive Function And Interoceptive Awareness In Heart Failure Outpatients. Circulation 2021;144:A9159-A9159.
- [Result] Salmoirago-Blotcher E, Walaska K, Trivedi D, Dunsiger S, Breault C, Levine D, Wu JR, Cohen R. Mind Your Heart: Exploring Feasibility, Acceptability, and Preliminary Effects of Phone-Delivered Mindfulness Training on Medication Adherence in Outpatients With Chronic Heart Failure. J Cardiovasc Nurs. 2022 Nov-Dec 01;37(6):595-602. doi: 10.1097/JCN.0000000000000891. Epub 2022 Jan 24. PMID 35067596

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mindfulness Training (MT)
Started | 33
Completed | 29
Not Completed | 4
Not completed — Death | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Mindfulness Training (MT): Eight, 30-minute phone delivered MT sessions once a week for 8 weeks
  Mindfulness Training (MT): Participants assigned to the MT condition will receive a phone-delivered 30-minute mindfulness training once a week for 8 weeks. In addition to the weekly training session, participants were instructed to practice mindfulness techniques for 20 minutes daily using a standardized audio recording to guide the participant through the techniques learned with the instructor.
Arm/Group | Mindfulness Training (MT)
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.3 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 23
  More than one race | 2
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Retention Rate
Description: Percentage of participants retained in the study (n enrolled/n retained X 100)
Time Frame: 3 months, 6 months
Population: 1 participant withdrew from the study and 1 died before the intervention started; these participants were not include in final analyses.
Measure: Count of Participants; unit: Participants
Groups:
- Mindfulness Training (MT): Eight, 30-minute phone delivered MT sessions once a week for 8 weeks
  Mindfulness Training (MT): Participants assigned to the MT condition will receive a phone-delivered 30-minute mindfulness training once a week for 8 weeks. In addition to the weekly training session, participants will be instructed to practice mindfulness techniques for 15 minutes daily using a standardized audio recording to guide the participant through the techniques learned with the instructor.
Arm/Group | Mindfulness Training (MT)
Number analyzed (Participants) | 31
Participants
  3 months | 31
  6 months | 29

2. Primary Outcome: Intervention Acceptability
Description: Self-reported intervention enjoyment scale (1 = did not enjoy to 5 = enjoyed very much). Scores range from 1 to 5; higher scores mean a better outcome. The metric for this study was the percentage of participants indicating high intervention enjoyment (a score of 5).
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Training (MT)
Number analyzed (Participants) | 31
Participants | 24

3. Secondary Outcome: Self-reported Medication Adherence
Description: The Voils extent of non-adherence scale ranges from 1-5. Higher scores represent greater non-adherence.
Time Frame: baseline, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training (MT)
Number analyzed (Participants) | 31
score on a scale
  Baseline | 2.8 (2.6)
  3 months | 2.6 (0.6)
  6 months | 2.6 (0.3)

4. Secondary Outcome: Objectively-assessed Medication Adherence
Description: Medication Event Monitoring Systems (MEMS). Proportion of medication taken/medication prescribed x 100, averaged over 30 days. Range is 0-100%. Lower values indicate worse adherence.
Time Frame: baseline, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: percentage of meds taken/prescrib
Arm/Group | Mindfulness Training (MT)
Number analyzed (Participants) | 31
percentage of meds taken/prescrib
  Baseline | 73 (28)
  3 months | 58 (35)
  6 months | 61 (37)

5. Secondary Outcome: Functional Capacity
Description: 6-min walk test (6MWT) distance. The 6 min walk test measures the distance a patient can walk on a level course in 6 min. It is a measure of functional capacity that correlates with peak oxygen uptake and is positively associated with survival in patients with cardiovascular disease. A higher value (in meters) indicates better functional capacity. The 6MWT distance in healthy adults has been reported to range from 400 to 700 meters.
Time Frame: baseline, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Mindfulness Training (MT)
Number analyzed (Participants) | 31
meters
  baseline | 350 (93)
  3 months | 378 (97)
  6 months | 374 (95)

6. Other Pre Specified Outcome: The Flanker Inhibitory Control and Attention Test
Description: Cognitive function was assessed using the NIH Toolbox Fluid Cognition Battery. Each neurocognitive test was independently completed by study participants (3-5 minutes each) using a study tablet after a baseline practice trial. For each cognitive measure we report age-adjusted scores, which are automatically generated by the NIH Toolbox software. For all measures, higher scores indicate better cognitive performance.
  The Flanker Inhibitory Control and Attention Test is a measure of executive function, attention and inhibitory control. Participants are instructed to focus on a stimulus while inhibiting attention to another stimulus (arrows). Sometimes the middle stimulus points in the same direction as the "flankers" (congruent) and sometimes in the opposite direction (incongruent) over 20 trials.
Time Frame: baseline, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training (MT)
Number analyzed (Participants) | 31
score on a scale
  Baseline | 87.9 (14.5)
  3 months | 93.2 (16.0)
  6 months | 92.6 (17.6)

7. Other Pre Specified Outcome: The Dimensional Change Card Sort Test
Description: The Dimensional Change Card Sort Test is a measure of cognitive flexibility and attention. Two target pictures are presented that vary along two dimensions (e.g., shape and color). Participants are asked to match a series of bivalent test pictures (e.g., yellow balls and blue trucks) to the target pictures, first according to one dimension (e.g., color) and then, after a number of trials, according to the other dimension (e.g., shape). The relevant dimension for sorting is indicated by a cue word (e.g., "shape" or "color") that appears on the screen for all participants. Age-adjusted scores are calculated automatically by the NIH Toolbox software. Higher scores indicate better function.
Time Frame: Baseline, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training (MT)
Number analyzed (Participants) | 31
score on a scale
  Baseline | 101 (19.7)
  3 months | 100.7 (10.0)
  6 months | 100.6 (20.1)

8. Other Pre Specified Outcome: Oral Symbol Digit Test
Description: The Oral Symbol digit test is a measure of working memory and processing speed. A key with nine abstract symbols is presented - each paired with a number between 1 and 9. Participants are asked to verbally indicate which numbers go with the symbols that are presented in a long string on the computer screen. The participant is given 120 seconds to call out as many numbers that go with the corresponding symbols as he/she can - in order, without skipping any. Age-adjusted scores were calculated automatically by the NIH Toolbox software. Higher scores indicate better function.
Time Frame: baseline, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training (MT)
Number analyzed (Participants) | 31
score on a scale
  Baseline | 58.8 (18.0)
  3 months | 65.7 (22.0)
  6 months | 62.8 (23.5)

9. Other Pre Specified Outcome: Picture Sequence Memory Test
Description: The Picture Sequence Memory Test is a measure of episodic memory. Sequences of pictured objects and activities are presented in a particular order. The participants are asked to reproduce the sequence of pictures that is shown on the screen. Participants respond by dragging pictures from the yellow box on the screen into the gray boxes on the screen.
  Age-adjusted scores were calculated automatically by the NIH Toolbox software. Higher scores indicate better function.
Time Frame: baseline, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training (MT)
Number analyzed (Participants) | 31
score on a scale
  Baseline | 98.2 (15.2)
  3 months | 102.1 (18.8)
  6 months | 109.9 (20.0)

10. Other Pre Specified Outcome: List Sorting Working Memory Test
Description: The List Sorting Working Memory Test is a measure of working memory. Pictures of foods and animals are displayed with accompanying audio recording and written text (e.g., "elephant"), and the participant is asked to say the items back in size order from smallest to largest, first within a single dimension (either animals or foods) and then on two dimensions (foods, then animals). Age-adjusted scores were calculated automatically by the NIH Toolbox software. Higher scores indicate better function.
Time Frame: baseline, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training (MT)
Number analyzed (Participants) | 31
score on a scale
  Baseline | 98.2 (13.7)
  3 months | 101.5 (14.9)
  6 months | 100.3 (62.8)

11. Other Pre Specified Outcome: Depressive Symptoms
Description: Hospital Anxiety and Depression Scale depression scores. Score range 0-21. Higher scores indicate greater psychological morbidity.
Time Frame: baseline, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Mindfulness Training (MT): Eight, 30-minute phone delivered MT sessions once a week for 8 weeks
  Mindfulness Training (MT): Participants assigned to the MT condition will receive a phone-delivered 30-minute mindfulness training once a week for 8 weeks. ). In addition to the weekly training session, participants will be instructed to practice mindfulness techniques for 20 minutes daily using a standardized audio recording to guide the participant through the techniques learned with the instructor.
Arm/Group | Mindfulness Training (MT)
Number analyzed (Participants) | 31
score on a scale
  Baseline | 3.6 (3.3)
  3 months | 4.3 (3.2)
  6 months | 4.9 (3.6)

12. Other Pre Specified Outcome: Sleep Quality
Description: Pittsburgh Sleep Quality Index. Self-report measure of sleep quality and quantity. Higher scores indicate better sleep quality and quantity. The overall score range is 0-21.
Time Frame: baseline, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training (MT)
Number analyzed (Participants) | 31
score on a scale
  baseline | 7.2 (3.9)
  3 months | 6.9 (3.9)
  6 months | 7.6 (4.6)

13. Other Pre Specified Outcome: Interoceptive Awareness: Noticing Score
Description: The Multidimensional Assessment of Interoceptive Awareness (MAIA) is a 32-item, self-report measure composed of eight individual scales, specifically: Noticing; Not Distracting; Not-Worrying; Attention Regulation; Emotional Awareness; Self-Regulation; Body Listening; and Trusting. Items are rated on a 6-point Likert scale (0-5) with '0' indicating 'Never' and '5' indicating 'Always'. For each subscale, items were summed; higher scores indicate higher levels of interoceptive awareness. This instrument has adequate to excellent internal-consistency reliability, with Cronbach's alphas between 0.66 and 0.87, and > 0.70 for five of the eight scales.
  The theoretical range for the noticing subscale score was 0-20.
Time Frame: baseline, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training (MT)
Number analyzed (Participants) | 31
score on a scale
  baseline | 12.7 (4.0)
  3 months | 14.5 (4.1)
  6 months | 15.0 (4.0)

14. Other Pre Specified Outcome: Interoceptive Awareness: Not Distracting Score
Description: The Multidimensional Assessment of Interoceptive Awareness (MAIA) is a 32-item, self-report measure composed of eight individual scales, specifically: Noticing; Not Distracting; Not-Worrying; Attention Regulation; Emotional Awareness; Self-Regulation; Body Listening; and Trusting. Items are rated on a 6-point Likert scale (0-5) with '0' indicating 'Never' and '5' indicating 'Always'. For each subscale, items were summed; higher scores indicate higher levels of interoceptive awareness. This instrument has adequate to excellent internal-consistency reliability, with Cronbach's alphas between 0.66 and 0.87, and > 0.70 for five of the eight scales.
  The theoretical range for the not distracting subscale score was 0-15.
Time Frame: baseline, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training (MT)
Number analyzed (Participants) | 31
score on a scale
  baseline | 6.6 (3.2)
  3 months | 7.2 (3.3)
  6 months | 7.3 (4.0)

15. Other Pre Specified Outcome: Interoceptive Awareness: Not Worrying Score
Description: The Multidimensional Assessment of Interoceptive Awareness (MAIA) is a 32-item, self-report measure composed of eight individual scales, specifically: Noticing; Not Distracting; Not-Worrying; Attention Regulation; Emotional Awareness; Self-Regulation; Body Listening; and Trusting. Items are rated on a 6-point Likert scale (0-5) with '0' indicating 'Never' and '5' indicating 'Always'. For each subscale, items were summed; higher scores indicate higher levels of interoceptive awareness. This instrument has adequate to excellent internal-consistency reliability, with Cronbach's alphas between 0.66 and 0.87, and > 0.70 for five of the eight scales.
  The theoretical range for the not-worrying subscale was 0-15.
Time Frame: baseline, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training (MT)
Number analyzed (Participants) | 31
score on a scale
  baseline | 8.2 (2.1)
  3 months | 8.3 (2.4)
  6 months | 7.8 (2.7)

16. Other Pre Specified Outcome: Interoceptive Awareness: Attention Regulation Score
Description: The Multidimensional Assessment of Interoceptive Awareness (MAIA) is a 32-item, self-report measure composed of eight individual scales, specifically: Noticing; Not Distracting; Not-Worrying; Attention Regulation; Emotional Awareness; Self-Regulation; Body Listening; and Trusting. Items are rated on a 6-point Likert scale (0-5) with '0' indicating 'Never' and '5' indicating 'Always'. For each subscale, items were summed; higher scores indicate higher levels of interoceptive awareness. This instrument has adequate to excellent internal-consistency reliability, with Cronbach's alphas between 0.66 and 0.87, and > 0.70 for five of the eight scales.
  The theoretical range for the attention regulation subscale score was 0-35.
Time Frame: baseline, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training (MT)
Number analyzed (Participants) | 31
score on a scale
  baseline | 20.1 (7.9)
  3 months | 24.2 (6.5)
  6 months | 23.5 (5.6)

17. Other Pre Specified Outcome: Interoceptive Awareness: Emotional Awareness Score
Description: The Multidimensional Assessment of Interoceptive Awareness (MAIA) is a 32-item, self-report measure composed of eight individual scales, specifically: Noticing; Not Distracting; Not-Worrying; Attention Regulation; Emotional Awareness; Self-Regulation; Body Listening; and Trusting. Items are rated on a 6-point Likert scale (0-5) with '0' indicating 'Never' and '5' indicating 'Always'. For each subscale, items were summed; higher scores indicate higher levels of interoceptive awareness. This instrument has adequate to excellent internal-consistency reliability, with Cronbach's alphas between 0.66 and 0.87, and > 0.70 for five of the eight scales.
  The theoretical range for the emotional awareness score was 0-25.
Time Frame: baseline, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training (MT)
Number analyzed (Participants) | 31
score on a scale
  baseline | 15.9 (5.2)
  3 months | 18.3 (5.3)
  6 months | 17.9 (5.3)

18. Other Pre Specified Outcome: Interoceptive Awareness: Self-regulation Score
Description: The Multidimensional Assessment of Interoceptive Awareness (MAIA) is a 32-item, self-report measure composed of eight individual scales, specifically: Noticing; Not Distracting; Not-Worrying; Attention Regulation; Emotional Awareness; Self-Regulation; Body Listening; and Trusting. Items are rated on a 6-point Likert scale (0-5) with '0' indicating 'Never' and '5' indicating 'Always'. For each subscale, items were summed; higher scores indicate higher levels of interoceptive awareness. This instrument has adequate to excellent internal-consistency reliability, with Cronbach's alphas between 0.66 and 0.87, and > 0.70 for five of the eight scales.
  The theoretical range for the self-regulation score was 0-20.
Time Frame: baseline, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training (MT)
Number analyzed (Participants) | 31
score on a scale
  baseline | 11.7 (5.0)
  3 months | 14.7 (3.6)
  6 months | 14.5 (3.9)

19. Other Pre Specified Outcome: Interoceptive Awareness: Body Listening Score
Description: The Multidimensional Assessment of Interoceptive Awareness (MAIA) is a 32-item, self-report measure composed of eight individual scales, specifically: Noticing; Not Distracting; Not-Worrying; Attention Regulation; Emotional Awareness; Self-Regulation; Body Listening; and Trusting. Items are rated on a 6-point Likert scale (0-5) with '0' indicating 'Never' and '5' indicating 'Always'. For each subscale, items were summed; higher scores indicate higher levels of interoceptive awareness. This instrument has adequate to excellent internal-consistency reliability, with Cronbach's alphas between 0.66 and 0.87, and > 0.70 for five of the eight scales.
  The theoretical range for the body listening score was 0-15.
Time Frame: baseline, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training (MT)
Number analyzed (Participants) | 31
score on a scale
  baseline | 7.4 (4.2)
  3 months | 8.9 (3.4)
  6 months | 9.6 (4.0)

20. Other Pre Specified Outcome: Interoceptive Awareness: Trusting Score
Description: The Multidimensional Assessment of Interoceptive Awareness (MAIA) is a 32-item, self-report measure composed of eight individual scales, specifically: Noticing; Not Distracting; Not-Worrying; Attention Regulation; Emotional Awareness; Self-Regulation; Body Listening; and Trusting. Items are rated on a 6-point Likert scale (0-5) with '0' indicating 'Never' and '5' indicating 'Always'. For each subscale, items were summed; higher scores indicate higher levels of interoceptive awareness. This instrument has adequate to excellent internal-consistency reliability, with Cronbach's alphas between 0.66 and 0.87, and > 0.70 for five of the eight scales.
  The theoretical range for the trusting subscale score was 0-15.
Time Frame: baseline, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training (MT)
Number analyzed (Participants) | 31
score on a scale
  baseline | 9.8 (3.9)
  3 months | 11.1 (2.8)
  6 months | 11.3 (3.5)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Mindfulness Training (MT)
All-Cause Mortality (participants affected / at risk) | 2/31
Serious Adverse Events (participants affected / at risk) | 3/31
Other Adverse Events (participants affected / at risk) | 8/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindfulness Training (MT) (N=31)
sudden cardiac death (Cardiac disorders) | 1 (1)
death (Cardiac disorders) | 1 (1)
stroke (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindfulness Training (MT) (N=31)
influenza (Infections and infestations) | 1 (1)
uncontrolled hypertension (Cardiac disorders) | 1 (1)
fall (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Impacted tooth (Surgical and medical procedures) | 1 (1)
pneumonia (Infections and infestations) | 1 (1)
car accident (Social circumstances) | 1 (1)
elective surgery (Surgical and medical procedures) | 1 (1)

LIMITATIONS AND CAVEATS:
This study did not accrue the planned number of participants (n=50) due the to Covid-19 pandemic leading to a smaller than planned sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT03571581/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/81/NCT03571581/ICF_001.pdf